CLINICAL TRIAL: NCT01271972
Title: A Phase 1 Study of REGN910 Administered Every 2 Weeks in Patients With Advanced Solid Malignancies
Brief Title: Study of Nesvacumab (REGN910/ SAR307746)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R910-ST-1010
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 (Experimental): Dose 1
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Cohort 2 (Experimental): Dose 2
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Cohort 3 (Experimental): Dose 3
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Cohort 4 (Experimental): Dose 4
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Cohort 5 (Experimental): Dose 5
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Expansion Cohort 1 (Experimental): Dose 4
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)
- Expansion Cohort 2 (Experimental): Dose 5
  Interventions: Drug: nesvacumab (REGN910/ SAR307746)

INTERVENTIONS:
Drug: nesvacumab (REGN910/ SAR307746)

SUMMARY:
This is an open-label, multicenter, ascending, multiple dose study of nesvacumab (REGN910/ SAR307746) administered IV every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of advanced solid malignancy.
2. ECOG performance status 0 - 1
3. Adequate hepatic, renal and bone marrow function
4. At least 3 weeks since last dose of chemotherapy, hormonal therapy or radiotherapy
5. At least 6 weeks since last dose of bevacizumab
6. At least 4 weeks since last surgery
7. At least 4 weeks since last dose of investigational treatment

Exclusion Criteria:

1. Patients with brain metastases, spinal cord compression, carcinomatous meningitis, or other evidence of central nervous system involvement
2. Patients with serious non healing wound or acute ulcer
3. Either systolic blood pressure >150 mm Hg or diastolic blood pressure >95 mm Hg
4. Patients with medical history of myocardial infarction, unstable angina pectoris, coronary/ peripheral artery bypass graft, congestive heart failure or ventricular arrhythmia
5. Patients with deep vein thrombosis or pulmonary embolism within last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerable dose or recommended phase 2 dose of nesvacumab (REGN910/ SAR307746) in patients with advanced solid malignancies | 28 days

SECONDARY OUTCOMES:
PK/PD profile | 28 days
Immunogenicity | 28 days
Anti-tumor activity | 28 days
Correlative biomarkers | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- United States (2):
  - San Francisco, California
  - San Antonio, Texas
- Toronto, Ontario, Canada